CLINICAL TRIAL: NCT03240770
Title: Effect of VPro5 Therapy on Clear Aligner Tracking: a Randomized Clinical Trial
Brief Title: Effect of VPro5 Therapy on Clear Aligner Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mani Alikhani (Industry)
Collaborators: Propel Orthodontics, LLC (Industry)
Responsible Party: Sponsor-Investigator, Mani Alikhani, Director, Consortium for Translational Orthodontic Research
Organization: Consortium for Translational Orthodontic Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VPro5 + Aligners
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Malocclusion
Keywords: HFV; HFA; High Frequency Vibration
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- 14 Day Tray + Sham (No Intervention): Trays worn at 14 day intervals + Sham
- 7 Day Tray + Sham (Experimental): Trays worn at 7 day intervals (Deviation from Standard Tray Wear Time (14 Days))
  + Sham
  Interventions: Other: Deviation from Standard Tray Wear Time (14 Days)
- 5 Day Tray + Sham (Experimental): Trays worn at 5 day intervals (Deviation from Standard Tray Wear Time (14 Days))
  + Sham
  Interventions: Other: Deviation from Standard Tray Wear Time (14 Days)
- 7 Day Tray + VPro5 (Experimental): Trays worn at 7 day intervals (Deviation from Standard Tray Wear Time (14 Days))
  + HFV with the VPro5 device at 5 min/day
  Interventions: Device: VPro5 device; Other: Deviation from Standard Tray Wear Time (14 Days)
- 5 Day Tray + VPro5 (Experimental): Trays worn at 5 day intervals (Deviation from Standard Tray Wear Time (14 Days))
  + HFV with the VPro5 device at 5 min/day
  Interventions: Device: VPro5 device; Other: Deviation from Standard Tray Wear Time (14 Days)

INTERVENTIONS:
Device: VPro5 device — Use of the VPro5 device for 5 minutes a day
  Arms: 5 Day Tray + VPro5; 7 Day Tray + VPro5
Other: Deviation from Standard Tray Wear Time (14 Days) — Patients reduced Tray Wear Time Interval (14 Days)
  Arms: 5 Day Tray + Sham; 5 Day Tray + VPro5; 7 Day Tray + Sham; 7 Day Tray + VPro5

SUMMARY:
The investigators hypothesize that brief, daily application of HFA will increase the efficiency of clear aligner treatment by altering PDL metabolism without increasing pain or discomfort. The investigators will divide subjects into 5 groups changing clear aligners at different time intervals with or without HFA application for 5 minutes/day to assess the effect on: time intervals between aligners, cytokine activity, and pain perception.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 - 45 years of age
2. Subject is willing and able to comply with all study procedures and sign Informed consent/HIPAA forms
3. Subject must have complete adult dentition (excluding third molars)
4. Subjects must have class I malocclusion or mild class II/III malocclusions
5. Subject is at least one month into aligner treatment.
6. Subject has history of and current healthy oral hygiene (PD is<4mm, GI<1, and PI=1)

Exclusion Criteria:

1. Subjects who have received periodontal treatment in the previous 6 months
2. Subjects who are taking medication that could affect the level of inflammation, such as chronic antibiotics, phenytoin, cyclosporin, ant-inflammatory drugs, systemic corticosteroids, or calcium channel blockers.
3. Subjects missing adult teeth (except the 3rd molars) or with severe class II or class III malocclusion.
4. Subjects with skeletal class I but extreme dental malocclusion
5. Severe crowding that require extraction
6. More than 4 mm positive overjet and more than 2 mm negative overjet
7. Extreme deep bite (more than 90%);
8. Severe openbite (more than 2 mm)
9. Pregnant women
10. Subjects do not have any systemic diseases effecting bone metabolism
11. Smoking
12. Vulnerable subjects per IRB definitions
13. Subjects with current caries
14. Subjects that require interproximal reduction or attachments during the study period
15. Subjects who are non-compliant regarding aligner wear or VPro5 recommended daily usage

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Average Aligner Tracking Percentage | Through study completion, average of 25 days
  Average assessed via measurement of intraoral scan and prediction software

SECONDARY OUTCOMES:
Cytokine Levels | Through study completion, average of 25 days
Pain Perception via Numerical Rating Scale | Day 1 and Day 3 of each aligner

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - CTOR, Hoboken, New Jersey
  - Orthodontia Studio, Hoboken, New Jersey
  - House of Orthodontia, Brooklyn, New York
  - Atique Orthodontics, San Antonio, Texas